CLINICAL TRIAL: NCT00810212
Title: A Prospective, Multicenter, Randomized, Open-Label, Controlled Study Evaluating Safety and Preliminary Efficacy of NeoFuse When Combined With Mastergraft Granules in Subjects Undergoing Posterolateral Lumbar Fusion With Instrumentation
Brief Title: Safety and Efficacy Study of NeoFuse in Subjects Requiring Posterolateral Lumbar Fusion
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor preferred a better study design
Sponsor: Mesoblast, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSB-SF002
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Degenerative Disc Disease; Degenerative Spondylolisthesis; Spinal Stenosis
Keywords: Degenerative disc disease; Spondylolisthesis; Spinal stenosis; Stem cell; Spinal Fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis; Spondylolisthesis | interventions — Transplantation, Autologous; Spinal Fusion

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of four (4) parallel treatment arms; autograft standard of care control, or one of three (3) doses of mesenchymal precursor cells (MPCs) combined with MasterGraft Granules. Subjects randomized to receive investigational product will be treated with one of the following three doses of allogeneic MPCs in 4 milliliters (mLs) per posterolateral lumbar fusion (PLF) level (204 mLs per side): 25 million (M), 50M or 75M MPCs per PLF level (or a total dose of 50 million, 100 million or 150 million MPCs if subject undergoes fusion at two levels). Each of the four treatment groups will include six (6) evaluable subjects.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Autograft
  Interventions: Procedure: PLF with autograft
- 2 (Experimental): Low Dose MPCs
  Interventions: Biological: PLF with NeoFuse
- 3 (Experimental): Medium Dose MPCs
  Interventions: Biological: PLF with NeoFuse
- 4 (Experimental): High Dose MPCs
  Interventions: Biological: PLF with NeoFuse

INTERVENTIONS:
Procedure: PLF with autograft — 6 subjects
  Other Names: spinal fusion
  Arms: 1
Biological: PLF with NeoFuse — 6 subjects low dose
  Other Names: spinal fusion; stem cell
  Arms: 2
Biological: PLF with NeoFuse — 6 subjects medium dose
  Other Names: spinal fusion; stem cell
  Arms: 3
Biological: PLF with NeoFuse — 6 subjects high dose
  Other Names: spinal fusion; stem cell
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate safety and preliminary efficacy of Neofusetm in subjects with a diagnosis of degenerative disc disease (DDD) in 1 or 2 adjacent vertebral levels between L1 and S1 and undergoing posterolateral lumbar fusion.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, open-label controlled Phase 1b/2a study designed to evaluate the safety and preliminary efficacy of MPCs combined with MasterGraft Granules when compared to use of autologous bone graft in the posterolateral fusion site in subjects requiring interbody fusion in combination with instrumented 1 or 2 level PLF procedure. All subjects in this study will undergo a 1 or 2-level (2 or 3 vertebrae) interbody fusion without the use of the investigational product.

In addition to the interbody fusion procedure, subjects will undergo an instrumented posterolateral fusion. NeoFuse plus MasterGraft Granules at one of three doses or autograft will be implanted in the posterolateral lumbar fusion site(s) only.

After the screening and surgical visits, each subject will be evaluated clinically and radiographically within 3 days and 30 days after surgery, and at 3, 6, 9, and 12 months after surgery.

Subjects will be evaluated at 24 and 36 months after surgery for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females at least 18 years of age, but not older than 70.
2. Have the ability to understand the requirements of the study, to provide written informed consent, and to comply with the study protocol.
3. Have the ability to understand and provide written authorization for the use and disclosure of personal health information (PHI) [per Health Insurance Portability and Accountability Act (HIPAA) privacy ruling in the US or applicable regulations outside the US].
4. Have a documented symptomatic diagnosis of DDD at L1-S1 with or without stenosis and with or without up to and including Grade II degenerative spondylolisthesis
5. Have clinical symptoms of neurogenic claudication.
6. Have failed 6 months of non-operative low back pain management.
7. Are candidates for lumbar interbody fusion with autograft in combination with posterolateral fusion and require surgery at a 1 or 2 adjacent vertebral levels between L1 and S1
8. Have a stable screening electrocardiogram (ECG), as determined by the investigator that would not preclude surgery -

Exclusion Criteria:

1. Female subjects who are pregnant or nursing, or women planning to become pregnant during the first year (12 months) following surgery.
2. Have a current or prior history within the last 3 years of neoplasm (excluding basal cell carcinoma) and/or any active neoplasm within the last 24 months, prior to screening.
3. Have osteoporosis as defined by a DEXA T score of ≤ -3.5 or a history of fragility fractures or other significant bone disease contraindicating the use of spinal instrumentation.
4. Have a documented medical history or radiographic evidence of a metabolic bone disease or other condition which would negatively impact the bone healing process.
5. Have a positive screen for human immunodeficiency virus (HIV) antibodies
6. Have had treatment with any investigational therapy or device within 6 months of study surgery and/or plans to participate in any other allogeneic stem cell/progenitor cell therapy trial during the 3-year follow-up period.
7. Have been a recipient of prior stem cell/progenitor cell therapy for spinal fusion surgery.
8. Have a body mass index (BMI) > 35.
9. Have 20% or greater anti-human leukocyte antigen (HLA) antibody titer and/or has antibody specificities to donor HLA antigens.
10. Are transient or has been treated in the last 6 months before enrollment for alcohol and/or drug abuse in an inpatient substance abuse program.

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of NeoFuse (allogeneic mesenchymal precursor cells [MPCs] when combined with MasterGraft Resorbable Ceramic granules as a carrier for posterolateral lumbar fusion (PLF) with instrumentation | 3 years

SECONDARY OUTCOMES:
To evaluate the overall fusion success with NeoFuse plus carrier compared to autograft using CT scans and x-ray of the involved lumbar spine levels and access the change in outcomes (ODI, SF-36) and pain (VAS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Donna Skerrett, MD, Principal Investigator — Mesoblast, Ltd., c/o Angioblast Systems, Inc.
Locations (1):
- Texas Back Institute, Plano, Texas, United States